CLINICAL TRIAL: NCT07333612
Title: Comparison of Immunoblotting Bands Pattern in Patients With Treated Versus Untreated Inactive Echinococcal Cysts of the Liver
Brief Title: IM Bands in Inactive Hepatic CE
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Raffaella Lissandrin, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: 08075323
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Cystic Echinococcosis
MeSH Terms: conditions — Echinococcosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
Comparison of immunoblotting bands pattern in patients with treated versus untreated echinococcal cysts of the liver

ELIGIBILITY:
Inclusion Criteria:

* Only Hepatic echinococcal cysts
* Age > 18 years
* At leat 2 clinical evaluation

Exclusion Criteria:

* different location of echinococcal cysts
* Age < 18 years --less then 2 clinical evalutation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients affected by cystic echinococcosis of the liver.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with spontaneously inactivated hepatic CE cysts with positive WB and RT t differente times from diagnosis. | from September 2024 to September 2026
  from 0 to 100%

SECONDARY OUTCOMES:
Percentage of cysts that remaine inactive after treatment or reactivate | from september 2024 to September 2026
  from 0 to 100%
Percentage of patients with inactivated cysts after treatment with positive WB results at different time point from the first observation of an inactive stage. | from September 2024 to September 2026
  from 0 to 100%

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, PV, Italy